CLINICAL TRIAL: NCT01605695
Title: Determination of the Normal Human Plasma Level of Inducible Nitric Oxide Synthase (iNOS) Using the PliNOSa Test
Brief Title: Normal Human Plasma Level of iNOS Study
Status: Completed | Type: Observational
Sponsor: Research & Diagnostic Antibodies (Industry)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dr. Robert Webber, President and Project PI, Research & Diagnostic Antibodies
Other Study IDs: RDAbs 12-002; 1RC3GM093717-01 (NIH)
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Normal Human Plasma Level of iNOS
Keywords: reference range; plasma; inducible nitric oxide synthase; iNOS; healthy adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — heparinized plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal healthy adults: The concentration of iNOS will be measured in plasma samples obtained at the time of blood donation from normal healthy adult humans

SUMMARY:
The discovery that inducible nitric oxide synthase (iNOS) circulates in people who are developing the sepsis pathology has provided an opportunity to develop a first-in-class diagnostic test for the onset of sepsis. This study is designed to determine the normal human plasma level of circulating iNOS as the initial reference level against which hospitalized patients at risk for the development of sepsis can be compared to ascertain if the patient is at risk for becoming septic based upon an elevated level of plasma iNOS.

DETAILED DESCRIPTION:
Infections in intensive care units (ICUs) and other hospital settings can be caused by different types of organisms, such as bacteria and fungi. Yearly, these infections cause at least 2 million patients in the USA to enter the early stages of the sepsis pathology (pre-sepsis) which will lead to more than 750,000 cases of sepsis that can deteriorate into life-threatening severe sepsis with organ dysfunction and septic shock with multiple organ failure and result in more than 250,000 deaths per year. At present, an accurate clinical lab test to predict the onset of the sepsis pathology does not exist. Thus, there is a large unmet clinical lab need for a test that can aid physicians in assessing the risk their hospitalized patients have for developing the sepsis pathology. A reliable test for predicting very early the onset of sepsis would be a major medical breakthrough. However, a reference level for normal healthy individuals is needed against which plasma levels can be compared for increased (or decreased) levels of iNOS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-79 years of age
* In generally good health

Exclusion Criteria:

* Cannot be a prisoner

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Reference values will be obtained from 100 plasma samples obtained from healthy normal humans collected prospectively under an IRB approved protocol and informed consent after blood donation for use in research. The 100 normal human plasma samples will be assayed using the PliNOSa test.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determination of the normal healthy human reference range for plasma iNOS | At time of blood donation
  The primary endpoint is the determination of the normal human plasma level of iNOS as the reference interval of the mean and it's 95% confidence interval. .

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Webber, Ph.D., Principal Investigator — Research & Diagnostic Antibodies
Locations (1):
- Research & Diagnostic Antibodies, North Las Vegas, Nevada, United States

REFERENCES:
- [Background] How to Define and Determine Reference Intervals in the Clinical Laboratory - Approved Guidelines, Second Edition, C28 A2, Vol 20, No. 3.